CLINICAL TRIAL: NCT07181408
Title: Assessment of the Impact of Functional Foods Enriched With Cricket and Pea Proteins on Perceived Satiety and Consumer Sensory Acceptance
Brief Title: Perceived Satiety and Consumer Sensory Acceptance of Functional Foods Enriched With Edible Insect and Plant Proteins
Acronym: NOODLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NOODLE
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: insect protein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cricket Flour-Enriched Snack (Experimental): savory snack enriched with 15% cricket flour
  Interventions: Other: Snack enriched with 15% cricket flour
- Pea Flour-Enriched Snack (Experimental): savory snack enriched with 15% pea flour
  Interventions: Other: Snack enriched with 15% pea flour.
- Control Snack (Wheat Flour-Based) (Placebo Comparator): conventional savory snack made of wheat flour.
  Interventions: Other: Wheat flour-based control snack

INTERVENTIONS:
Other: Wheat flour-based control snack — Consumption of a single 50-gram portion of a wheat flour-based control snack.
  Arms: Control Snack (Wheat Flour-Based)
Other: Snack enriched with 15% cricket flour — Consumption of a single 50-gram portion of a snack enriched with 15% cricket flour (Acheta domesticus).
  Arms: Cricket Flour-Enriched Snack
Other: Snack enriched with 15% pea flour. — Consumption of a single 50-gram portion of a snack enriched with 15% pea flour.
  Arms: Pea Flour-Enriched Snack

SUMMARY:
This randomized, single-blind, triple crossover study investigated the effects of baked snacks containing either cricket flour (Acheta domesticus), pea flour (both at 15%), or a wheat flour-based control. One hundred adult participants were recruited and consumed each of the three products across separate sessions. Data were collected on sociodemographic characteristics, hunger and satiety perceptions using visual analogue scales (VAS), gastrointestinal tolerability via a post-consumption questionnaire, hedonic liking assessed with a 9-point scale, and sensory and emotional responses using Check-All-That-Apply (CATA) questionnaires.

DETAILED DESCRIPTION:
The present experimental study aimed to evaluate the subjective responses of consumers following the consumption of three types of savory snacks differing in protein composition: a conventional control snack, one enriched with cricket flour (Acheta domesticus), and one enriched with pea flour. The trial was designed as a randomized, single-blind, triple crossover intervention study. A total of 100 healthy adult volunteers were recruited, aged between 18 and 65 years, with a body mass index (BMI) ranging from 18.5 to 29.9 kg/m². Each participant consumed a single 50-gram portion of each product, with a seven-day washout period between sessions. The order of product administration was randomized. All tastings were carried out in a fasting state, preferably in the morning, to standardize metabolic conditions. During each session, the following data were collected:

* Sociodemographic characteristics, assessed at baseline via questionnaire;
* Perceived satiety, measured using a Visual Analogue Scale (VAS) at 60, 120, 180, 240, and 300 minutes after the end of the meal;
* Gastrointestinal tolerability, evaluated through a post-consumption questionnaire addressing symptoms such as bloating, nausea, and abdominal discomfort;
* Hedonic evaluation, assessed using a 9-point hedonic scale to determine product acceptability;
* Sensory and emotional responses, collected through Check-All-That-Apply (CATA) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer subjects aged between 18 and 65 years;
* Body mass index (BMI) between 18.5 and 29.9 kg/m²

Exclusion Criteria:

* Diagnosis of diabetes mellitus;
* Thyroid disorders;
* Food allergies;
* Gastrointestinal and/or systemic diseases (including renal, hepatic, cardiovascular, or any other organ-related conditions);
* Regular use of medications or dietary supplements;
* Pregnancy or lactation;
* Following specific dietary regimens (vegetarian or vegan).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Postprandial Subjective Satiety Perception | 60, 120, 180, 240, and 300 minutes post-consumption.
  Satiety perception will be assessed using the Visual Analogue Scale (VAS; 0-100 mm), where 0 = "not satiated at all" and 100 = "extremely satiated". Higher scores indicate greater satiety.
Postprandial Hunger | 60, 120, 180, 240, and 300 minutes post-consumption.
  Hunger perception will be assessed using the Visual Analogue Scale (VAS; 0-100 mm), where 0 = "not hungry at all" and 100 = "extremely hungry". Higher scores indicate greater hunger.
Postprandial Gastric Fullness | 60, 120, 180, 240, and 300 minutes post-consumption.
  Gastric fullness perception will be assessed using the Visual Analogue Scale (VAS; 0-100 mm), where 0 = "not full at all" and 100 = "extremely full". Higher scores indicate greater fullness.
Prospective Food Consumption | 60, 120, 180, 240, and 300 minutes post-consumption.
  Prospective food consumption will be assessed using the Visual Analogue Scale (VAS; 0-100 mm), where 0 = "no desire to eat at all" and 100 = "extreme desire to eat". Higher scores indicate greater desire for food intake.

SECONDARY OUTCOMES:
Gastrointestinal Symptoms Evaluation | Within 24 hours after snack intake.
  Self-reported evaluation of gastrointestinal symptoms potentially related to snack consumption, assessed using the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS uses a 10-point Likert scale (1 = no symptoms, 10 = very severe symptoms). Higher scores indicate more severe gastrointestinal symptoms.
Sensory Acceptability | Immediately after snack consumption.
  Evaluation of overall sensory acceptability of the snack products, including visual appearance, odor, taste, texture, general liking, and purchase intent. Assessments will be performed using a Visual Analogue Scale (VAS; 0-100 mm), where 0 mm represents "dislike extremely / not acceptable at all" and 100 mm represents "like extremely / highly acceptable". Higher scores indicate greater sensory acceptability.
Emotional and Descriptive Food Experience | Immediately after snack consumption.
  Exploration of the emotional and sensory descriptive dimension of the eating experience using Check-All-That-Apply (CATA) questionnaires. Participants will select all terms that describe their experience of the snack. Since this is a categorical measure, no numerical scale is applied. Data will be analyzed as the frequency of selection of each descriptor.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT07181408/Prot_ICF_000.pdf